CLINICAL TRIAL: NCT06510296
Title: Digital Mind Body Intervention Among Black and Hispanic Patients Living With Inflammatory Bowel Disease
Acronym: DMBI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-16064; 1K12TR004411 (NIH)
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Crohn's Disease; Ulcerative Colitis; Inflammatory Bowel Diseases
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Mind Body Intervention (Experimental): Participants randomized to the Digital Mind Body mobile intervention will receive a unique user identification (user ID) to access the DMBI mobile application. Randomized in a 2:1 ratio for DMBI intervention vs Waitlist Control
  Interventions: Behavioral: Digital Mind Body Intervention mobile application
- Waitlist Control (No Intervention): Patients randomized to the Waitlist Control arm/group will not receive the DMBI until the end of the study. During the study, to control for expectancy and attention, the Waitlist Control will receive a weekly email with generic tips on a healthy lifestyle in IBD. Randomized in a 2:1 ratio for DMBI intervention vs Waitlist Control

INTERVENTIONS:
Behavioral: Digital Mind Body Intervention mobile application — A DMBI mobile application with psychoeducation and skill-building in illness perception, coping, mindfulness, and disease acceptance informed by needs/barriers of Black and Hispanic patients with IBD who have elevated psychological distress and GI professionals caring for IBD patients.
  Arms: Digital Mind Body Intervention

SUMMARY:
The bidirectional effects between psychological distress and inflammatory bowel disease (IBD) activity mean that not only does increased IBD activity trigger psychological distress, but psychological distress triggers increased IBD activity (i.e., gut-brain interaction). Comorbid psychological distress is linked to increased health resource utilization and poor health-related quality of life (HRQoL). This has prompted calls for integrating psychological care into IBD practice with restoration of quality of life as a clinical target of IBD management alongside endoscopic healing. The IBD Social Cognitive Model (IBD SCM) posits that patient psycho-behavioral modifiers contribute to IBD outcomes and not disease modifiers alone. While a co-localized gastro-psychologist in an IBD medical home is an emerging mode of delivering psycho-behavioral care among people living with IBD, access and scalability of this form of support is not yet widespread, particularly in resource-limited settings. Though many people with IBD have significant psychological distress, mental health care is underutilized with cost cited as a barrier.

The emergence of digital interventions in clinical practice presents an opportunity to address access, scalability, and cost barriers. However, current testing of digital interventions to address gut-brain interactions (digital mind-body intervention, DMBI) among people with IBD involves mostly women with high educational attainment who have full time employment and do not receive social service benefits. Individuals with limited resources and those from racial and ethnic minority groups (e.g. Black, Hispanic) often have socioecological factors, such as healthcare access and mental health stigma, that impede their use of psycho-behavioral resources. DMBI development informed by participatory research approaches are, therefore, critical to facilitate equitable engagement and utilization. Beneficial effects of psycho-behavioral treatment among people with IBD are strongest for those who have psychological distress and for acceptance, mindfulness, and values-based approaches.

Although high quality evidence demonstrates psychological improvement with DMBI in IBD, feasibility and acceptability of applying DMBI to IBD patients from racial and ethnic minority groups is lacking.

DETAILED DESCRIPTION:
Prior to conducting the randomized pilot study, as part of Aim 1, patient focus groups will be conducted, based on the IBD social-cognitive model (IBD SCM), with a prototype DMBI to assess resonance and preferences on how to convey and display intervention concepts and components. Semi-structured interviews will be conducted among gastroenterology professionals (GIs) to assess perceived needs and barriers to DMBI acceptance and use in clinical care of Black and Hispanic patients with IBD, and define intervention elements.

Aim 2 will be guided by the needs/barriers identified in Aim 1, a functional DMBI app will be developed. A formative/summative evaluation of the app intervention will be conducted through iterative patient user testing to ensure functionality and usability (e.g. accessibility/ease of use, relevant and non-stigmatizing content).

Aim 3, the basis for this registration, will consist of an 8-week pilot of the refined DMBI intervention, developed in Aim 2 among a separate group of patients, to assess the feasibility and acceptability of DMBI among Black and Hispanic patients with IBD. It is anticipated that Aim 3 will not initiate until July, 2027. Earlier Aims, not represented in this record, are in progress.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* self-identify as Black/African American and/or Hispanic/Latino(a/x)
* diagnosed with Crohn's disease or ulcerative colitis
* ability to provide informed consent in English
* elevated psychological distress: at least one T-score within 2.5 standard deviations above the mean -- NIH Toolbox Perceived Stress Scale or in the domains of either Anxiety or Depression on the NIH PROMIS-29.

Exclusion Criteria:

* Anxiety, depression, or perceived stress T-scores above 2.5 standard deviations above the mean.
* Current suicidality, past suicide attempt, or psychiatric hospitalization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-07 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Feasibility - DMBI recruitment rate | 8 weeks
  DMBI recruitment rate will be determined by the proportion of eligible patients who enroll into the trial. A benchmark to define this feasibility outcome will be ≥ 30% of eligible patients enrolling.
Feasibility - DMBI retention rate | 8 weeks
  DMBI Retention rate will be determined by the proportion of enrolled patients who complete all DMBI modules. A benchmark to define this feasibility outcome will be ≥ 70% of enrolled patients completing all DMBI modules.
Feasibility - DMBI adherence | 8 weeks
  DMBI adherence will be assessed by the percentage of completed activities per module will be determined. A benchmark to define this feasibility outcome will be ≥ 50% of completed activities per module.

SECONDARY OUTCOMES:
Illness Perception | Week 0 (Baseline) and at 8 weeks
  The 8-item Brief Illness Perception Questionnaire (BIPQ) will be used to assess self-reported Illness Perception. Responses to the eight questions related are scored from 0 (negligible illness impact) to 10 (intense illness impact) for a possible scoring range of 0-80. Higher scores indicate more severe patient perception of illness impact. Group mean scores will be summarized.
IBD self-efficacy | Week 0 (Baseline) and at 8 weeks
  IBD self-efficacy will be evaluated based on the 13-item IBD Self Efficacy Scale (IBD-SES) which measure the composite score across four domains of self-efficacy (managing stress and emotions, medical care, symptoms and disease, and maintaining remission). Responses to the 13 questions are scored from 0 (Not sure at all) to 10 (Totally sure) for a possible scoring range of 0-130. Higher scores are associated with increased patient self-efficacy across the four domains. Group mean scores will be summarized.
Disease acceptance | Week 0 (Baseline) and at 8 weeks
  Patient disease acceptance will be assessed using the 20-item Digestive Disease Acceptance Questionnaire (DDAQ). The DDAQ consists of 20 statements asking patients to rate the truth of each statement on a scale ranging from 0 (Never True) to 6 (Always True) for an overall possible scoring range of 0-120. Higher scores are associated with increased patient disease acceptance. Group mean scores will be summarized.
Mindfulness | Week 0 (Baseline) and at 8 weeks
  Mindfulness is evaluated based on the 15-item Five Facet Mindfulness Questionnaire (FFMQ-15). The FFMQ measures mindfulness with regards to thoughts, experiences, and actions in daily life across five subscales. Responses to the positively worded statements (Statements 1-2, 5-6, 10-12, 15) are scored from 1 (Never or very rarely true) to 5 (Very often or always true). Responses to the negatively worded statements (Statements 3-4, 7-9, 13-14) are scored from 5 (Never or very rarely true) to 1 (Very often or always true) for an overall possible scoring range of 15-75. Higher scores are indicative of someone who is more mindful in their everyday life. Group mean scores will be summarized.
GI-specific symptom anxiety (GSA) | Week 0 (Baseline) and at 8 weeks
  GI-specific symptom anxiety will be based on responses to the 15-item Visceral Sensitivity Index (VSI) questionnaire. The VSI consists of 15 statements describing how people respond to abdominal symptoms/discomfort. Individual responses are scored on a scale ranging from 1 (Strongly Disagree) to 6 (Strongly Agree) yielding a range of possible scores from 15 (no GSA) to 90 (severe GSA). Lower scores are associated with higher GSA. Group mean scores will be summarized.
Resilience | Week 0 (Baseline) and at 8 weeks
  Resilience will be determined based on the 14-item Resilience Scale for Inflammatory Bowel Disease (RISE IBD) scale. RISE-IBD consists of 14 statements governing four domains scored on a scale ranging from 0-4. Positively worded statements in the survey (Statements 1-2, 4-5, 7, 9-13) are scored from 0 (Not True) to 4 (Always True) and negatively worded statements in the survey (Statements 3, 6, 8 and 14) are reverse scored from 0 (Always True) to 4 (Not True) for a possible overall scoring range of 0-56. Higher scores reflect greater patient resilience. Group mean scores will be summarized.
Health-related Quality of Life | Week 0 (Baseline) and at 8 weeks
  The Patient-Reported Outcomes Measurement Information System (PROMIS)-29 questionnaire will be used to assess Health-related Quality of Life. PROMIS-29 consists of 29 questions/statements which include 4 items across 7 domains along with a single Pain Intensity item. Pain Intensity is measured on a scale from 0 (No Pain) to 10 (Worst pain imaginable). Responses to the other 28 items are scored from 1-5. Raw scores are converted to a T-score that centers at mean T-score of 50 with a Standard Deviation of 10 in a general, reference population. Higher scores indicate higher degree of the measured trait. Group mean scores will be summarized.
IBD Activity for Crohn's Disease (CD) Patients | Week 0 (Baseline) and at 8 weeks
  For patients with CD, IBD activity will be assessed using the Short Crohn's Disease Activity Index (CDAI). The CDAI consists of 3 questions assessing CD symptoms/activity daily over the prior 7 days. The three questions relate to the number of liquid or soft stools each day; abdominal pain severity each day; and general well-being each day. Scoring is summarized as follows:
  44 + (2 x the number of liquid or soft stools each day for 7 days) + 5 x the sum of seven daily abdominal pain ratings (0 = none, 1 = mild, 2 = moderate, 3 = severe)] + 7 x the sum of seven general well-being ratings (0 = generally well, 1 = slightly under par, 2 = poor, 3 = very poor, 4 = terrible)]
  Overall CDAI scores range from 0 to approximately 600. Higher scores are associated with increased Crohn's disease severity. Group mean scores will be summarized.
IBD Activity for Ulcerative Colitis (UC) Patients | Week 0 (Baseline) and at 8 weeks
  For patients with UC, IBD activity will be assessed using Simple Clinical Colitis Activity index (SCCAI). The SCCAI consists of 6 questions assessing UC disease symptoms. Three questions: Bowel Frequency (per day), Urgency of Defecation, and Blood in Stool are scored on a 0-3 scale with higher scores indicating increasing severity). Bowel Frequency (per night) is scored from 0-2 with higher scores denoting greater frequency and General well-being is scored from 0-4 with higher scores indicative of decreasing well being. A final question assigns a point per extracolonic manifestation for any of the following features (uveitis, pyoderma gangrenosum, erythema nodosum, or arthropathy). Overall SCCAI range is 0-19 with higher overall scores being associated with increased severity of UC symptoms. Group mean scores will be summarized.

OTHER OUTCOMES:
Fecal Calprotectin Concentrations | Week 0 (Baseline) and at 8 weeks
  Stool samples will be collected at baseline and 8 weeks to measure fecal calprotectin levels. Stool samples will be analyzed using ELISA or an immunochromatographic assay. Reference rages vary but concentrations between 50-120 ug/g are considered moderate/borderline. Fecal Calprotectin concentrations greater than 120 ug/g are considered high/abnormal. Group mean fecal calprotectin concentrations will be summarized. Fecal calprotectin can be a surrogate marker for IBD. High levels of fecal calprotectin are indicative of intestinal inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Ruby Greywoode, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No